CLINICAL TRIAL: NCT07253103
Title: "Effects of a Resistance Physical Exercise Program in Multiple Myeloma Patients: A Randomized Controlled Trial Study Protocol".
Brief Title: Effects of a Resistance Physical Exercise Program in Multiple Myeloma Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, CARLOS MARTIN SANCHEZ, Director, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ExerciseMM2025
Record Dates: First submitted 2025-11-16; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma (MM); Exercise; Cancer
Keywords: Cancer; Exercise; Múltiple Myeloma; Physiotherapy; Protocol; Resistance
MeSH Terms: conditions — Multiple Myeloma; Motor Activity; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given the study design, it will not be possible to blind participants or assessors to the intervention. However, in order to preserve the objectivity of the results, the statistical analysis will be performed by an independent statistician who is not involved in the study and is unaware of the allocation of participants to the different groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Supervised physical exercise program
  Interventions: Other: Supervised physical exercise; Other: Home-based physical exercise program
- Control group (Experimental): Home-based physical exercise program
  Interventions: Other: Home-based physical exercise program

INTERVENTIONS:
Other: Supervised physical exercise — Participants will follow a supervised physical exercise program for 12 weeks.
  Arms: Intervention group
Other: Home-based physical exercise program — Participants will follow a home-based physical exercise program for 12 weeks.

SUMMARY:
The goal of this clinical trial is to learn if physical exercise improves quality of life, frailty and mental health in patients with multiple myeloma. It will also learn about the safety and adherence of the program. The main questions it aims to answer are:

Does physical exercise improves quality of life in patients with multiple myeloma? Does physical exercise improves frailty and mental health in patients with multiple myeloma? Researchers will compare supervised physical exercise and home-based unsupervised physical exercise.

Participants will:

Participate in one of the exercise programs, supervised or home-based, for 12 weeks. They will be completely evaluated before and after the intervention.

DETAILED DESCRIPTION:
Participants will be patients diagnosed with multiple myeloma (MM) who are undergoing active treatment and who will be recruited from the Haematology Department of Salamanca University Hospital.

Intervention The physical exercise programme has been specifically designed for people diagnosed with MM undergoing active treatment. To ensure methodological quality and reproducibility of the intervention, the recommendations of the Consensus on Exercise Reporting Template (CERT) [X] will be followed, a detailed description of which is included in the supplementary material (Table S2).

The programme will focus primarily on resistance training, supplemented by daily aerobic activities, and will last for a total of twelve weeks. The sample will be randomly assigned to two groups: an intervention group (IG) and a control group (CG), as described below.

1. Intervention group The IG will participate in a supervised resistance training programme, with two sessions per week, 12 weeks, supplemented by a home-based physical activity promotion programme to be carried out four times per week. All supervised sessions will be led by a physiotherapist at a health centre.
2. Control group The CG will only perform the home-based physical activity promotion program 4 days/week.

The randomisation process for this clinical trial will be carried out using Microsoft Excel 2020, which will generate a list of random numbers for the allocation of participants. Each participant will be assigned a unique number from this list: those with odd numbers will be assigned to the experimental group, and those with even numbers to the control group. This procedure ensures a random and balanced distribution between the groups, minimising possible biases and increasing the validity of the study results. Randomisation will be carried out by a member of staff from the Haematology Department of the University Hospital of Salamanca who will not be involved in the research.

Given the study design, it will not be possible to blind participants or assessors to the intervention. However, in order to preserve the objectivity of the results, the statistical analysis will be performed by an independent statistician who is not involved in the study and is unaware of the allocation of participants to the different groups.

For descriptive analysis, data normality will be asessed using the Kolmogorov-Smirnov and Shapiro-Wilk tests (the latter applicable in samples with n < 30). Variables with a normal distribution will be described using mean, standard deviation and range, while those that do not follow a normal distribution will be represented using median and interquartile range. Qualitative variables will be expressed in absolute frequencies and percentages.

In quantitative analysis, Pearson's correlation coefficient will be used to verify the validity of the assessment procedures used in the study, and Cronbach's alpha will be used to determine their internal reliability.

For comparisons between two means, the following will be applied: Student's t-test for independent samples (parametric), Mann-Whitney U test (non-parametric for independent samples), and Wilcoxon test (non-parametric for paired data). When comparing three or more means, an ANOVA for independent groups (parametric test with Snedecor's F test) will be used or, failing that, the Kruskal-Wallis test (non-parametric). In the case of repeated measures, Snedecor's F test will be applied for parametric data and Friedman's test for non-parametric data. Correlations will be analysed using Pearson's coefficient when the data follow a normal distribution and Spearman's coefficient when they do not. To identify the variables associated with the results of interest, a multivariate logistic regression analysis will be performed, including in the model those variables that are significant in the bivariate analysis or that are considered relevant to the study. For qualitative or categorical variables, contingency tables and the Chi-square test will be used in comparisons between two independent samples. A p-value < 0.05 will be considered significant, corresponding to a 95% confidence interval. All statistical analyses will be performed using IBM SPSS Statistics, version 28.0.1.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of MM undergoing active treatment.
* No regular physical activity during the previous eight weeks.
* Functional status (ECOG) 0-1.
* Signature of informed consent.

Exclusion criteria:

* Presence of medical contraindications for physical exercise, such as severe musculoskeletal disorders, severe cardiovascular disease, bone metastases, or other conditions that the medical team considers inappropriate.
* Inability to complete the initial assessment tests or difficulty performing basic exercises.
* Any other circumstance that, in the opinion of the investigators, may interfere with the objectives or conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | 12 weeks
  The primary outcome measure will be health related quality of life. Quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ). Specifically, the EORTC QLQ-C30 will be used, which is widely used to assess quality of life in cancer patients [X]. This instrument consists of 30 items, 24 of which are grouped into five functional domains: physical, role, emotional, cognitive, and social. It also includes three symptom scales-fatigue, pain, and nausea/vomiting-and an overall health status scale. Six other items assess additional symptoms such as dyspnoea, loss of appetite, insomnia, constipation, diarrhoea, and financial difficulties. Responses are recorded on a four-point scale ('none,' 'a little,' 'quite a bit,' 'a lot'), except for the general health and quality of life scales, which use a seven-point format. On the functional and overall health scales, higher scores indicate better health, while on the

SECONDARY OUTCOMES:
Frailty | 12 weeks
  Frailty will be assessed using the Short Physical Performance Battery (SPPB) scale [X], which comprises three components: a balance test, a gait speed test, and a chair rise test. The maximum possible score is 12 points, with higher scores reflecting a better level of physical function.
Anxiety and depression | 12 weeks
  The presence of anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS), a validated questionnaire widely used in different populations [X]. The scale consists of 14 items: seven corresponding to the anxiety subscale (HADS-A) and seven to the depression subscale (HADS-D). Each item is scored from 0 to 3, with separate scores obtained for both emotional dimensions.
Fatigue | 12 weeks
  Fatigue will be measured using the Functional Assessment of Cancer Therapy-Fatigue (FACT-F) subscale [X], a self-reported instrument designed to assess the severity of fatigue in cancer patients [X,X]. This widely used tool combines the 27 items of the FACT-General with 13 additional fatigue-specific items, generating a total score range between 0 and 160. Higher scores indicate lower perceived fatigue levels.
Sleep quality | 12 weeks
  Sleep quality will be assessed using the Athens Insomnia Scale (AIS), an eight-item self-administered scale developed by Soldatos [X] and validated for use in the Spanish population [X]. The first five items assess sleep disturbances-sleep onset, night-time awakenings, early awakening, total sleep duration, and overall quality-corresponding to criterion 'A' for the diagnosis of insomnia according to the ICD-10 classification. The remaining three items assess daytime consequences (well-being, physical and mental functioning, and daytime sleepiness), aligned with criterion 'C' of the same classification.
  Each item is scored on a Likert scale from 0 ('no problem') to 3 ('significant problem'), yielding a total range of 0 to 24. Higher scores indicate greater sleep disturbance, and values equal to or greater than 6 are considered indicative of clinically relevant insomnia [X].
Physical activity | 12 weeks
  The overall level of physical activity will be determined using the Spanish version of the International Physical Activity Questionnaire (IPAQ) [X]. This questionnaire consists of seven questions that assess the duration and frequency of physical activities of varying intensity:
  * Light activity (<600 MET-minutes/week), such as walking at home, at work or during leisure time.
  * Moderate activity (600-3000 MET-minutes/week), such as cycling, playing tennis or carrying light objects.
  * Vigorous activity (>3000 MET-minutes/week), which includes intense exercises such as aerobics, digging or weightlifting.
  The IPAQ also records the amount of time spent being inactive during the past week, providing a comprehensive overview of the participant's activity levels. The total physical activity score is calculated by adding up the vigorous, moderate and light activities expressed in MET-minutes/week [X].
Body composition | 12 weeks
  Various variables related to the participants' body composition will be collected. Height will be measured using a height gauge, and the rest of the parameters will be obtained by electrical bioimpedance, using the TANITA BC-418® device. The variables will include total body weight and appendicular muscle mass (ASM), defined as the sum of the muscle mass of the limbs. To calculate the appendicular muscle mass index (ASMI), the height-adjusted formula (AMM/height²) will be applied [X].
  Parameters such as visceral fat, body fat percentage (BF%), and body mass index (BMI) will also be assessed. To ensure the accuracy of the measurements, all participants will be weighed wearing minimal clothing and barefoot, thus reducing variability and ensuring that the results reliably reflect actual body composition [X].
Strength | 12 weeks
  The strength of the upper and lower limbs will be assessed using different procedures. For handgrip strength, the Jamar® hydraulic dynamometer (J00105, Lafayette Instrument Company, USA) will be used, which is considered the gold standard for this type of measurement [X]. Both hands will be assessed following the Southampton Protocol [X]. The participant will sit in a chair with a backrest, with the shoulder adducted and in neutral rotation, the elbow flexed at 90°, the forearm in a neutral position and the wrist in slight extension (0°-30°).
  Three consecutive measurements will be taken on each hand, with 5-second contractions and 10-second breaks between them. During the test, the participant will be encouraged to exert maximum effort. The second position of the dynamometer will be used in all cases, except for small hands, where the first position will be used (duly recorded). The same evaluator will perform all measurements, and the average or maximum value for each hand will be co
Physical performance | 12 weeks
  In addition to the SPPB, physical performance will be assessed using the four-metre walk test (4MWT), a complementary indicator of frailty. The participant will begin walking one metre before the starting line, where the stopwatch will be started, and will continue at their usual speed until four metres beyond the finish line. The test will be repeated three times and the best time achieved will be recorded

IPD SHARING:
Plan to Share IPD: Undecided
The datasets [GENERATED/ANALYZED] for this study can be found in the [NAME OF REPOSITORY] [LINK]. Please see the "Availability of data" section of Materials and data policies in the Author guidelines for more details.

REFERENCES:
- [Background] Fairman CM, Zourdos MC, Helms ER, Focht BC. A Scientific Rationale to Improve Resistance Training Prescription in Exercise Oncology. Sports Med. 2017 Aug;47(8):1457-1465. doi: 10.1007/s40279-017-0673-7. PMID 28074412
- [Background] Kirkham AA, Eves ND, Shave RE, Bland KA, Bovard J, Gelmon KA, Virani SA, McKenzie DC, Stohr EJ, Waburton DER, Campbell KL. The effect of an aerobic exercise bout 24 h prior to each doxorubicin treatment for breast cancer on markers of cardiotoxicity and treatment symptoms: a RCT. Breast Cancer Res Treat. 2018 Feb;167(3):719-729. doi: 10.1007/s10549-017-4554-4. Epub 2017 Nov 6. PMID 29110150